CLINICAL TRIAL: NCT03004443
Title: Inflammation-Induced CNS Glutamate Changes in Depression
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was suspended in March 2020 due to the COVID-19 pandemic and ultimately was terminated as it is not safe to test a potent anti-inflammatory drug with ongoing surges of COVID-19.
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Andrew H Miller, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00090667; 1R01MH112076-01 (NIH)
Record Dates: First submitted 2016-12-08; First posted 2016-12-28 (Estimated); Results first posted 2023-06-07 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Depression
Keywords: Psychiatry
MeSH Terms: conditions — Depression | interventions — Infliximab; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Infliximab (Experimental): Participants will be randomized to receive one intravenous (IV) infusion of infliximab.
  Interventions: Drug: Infliximab
- Placebo (Placebo Comparator): Participants will be randomized to receive one intravenous (IV) infusion of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Infliximab — Infliximab will be administered intravenously (IV) as 5 mg/kg body weight over a 2 to 2.5 hour period.
  Other Names: Remicade
  Arms: Infliximab
Drug: Placebo — Saline solution will be administered intravenously over a 2 to 2.5 hour period.
  Other Names: Saline solution
  Arms: Placebo

SUMMARY:
Increased inflammation has been implicated in the pathophysiology of a number of neuropsychiatric illnesses including mood disorders, which affect almost 30 million adults in the United States alone. One mechanism by which inflammation may alter behavior is through increasing brain glutamate, a neurotransmitter that in excess has been implicated in neuronal toxicity and resistance to conventional antidepressant therapy. The goal of the proposed research is to test the hypothesis that inflammation alters behavior through increasing glutamate in specific brain regions, ultimately leading to behavioral changes.

The proposed research is designed to determine the cause and effect relationship between inflammation and CNS glutamate as well as the relationship between CNS glutamate and specific symptoms. To accomplish these aims, investigators will administer a single infusion of either the tumor necrosis factor (TNF) antagonist infliximab or placebo (n=30 per group) to patients with high inflammation (CRP>3mg/L). A CRP>3mg/L was chosen because it is considered high inflammation according to guidelines by the American Heart Association. Moreover, a CRP>3mg/L is associated with significantly increased basal ganglia glutamate and with a clinical response to infliximab. Inflammatory biomarkers, basal ganglia glutamate as measured by MRS, and motivation and psychomotor activity will be assessed at baseline and days 1 and 3 and weeks 1 and 2 following infliximab or placebo administration.

DETAILED DESCRIPTION:
This study aims to test the hypothesis that increased inflammation causes increased basal ganglia glutamate and consequently anhedonia and psychomotor retardation in patients with major depressive disorder (MDD). Excessive inflammation and glutamate excitotoxicity are two pathways that have received increasing attention regarding the pathophysiology of neuropsychiatric disease including mood disorders. Patients with depression exhibit increased peripheral and central nervous system (CNS) markers of inflammation as well as altered CNS glutamate as measured by magnetic resonance spectroscopy (MRS). In addition, drugs that block either inflammation or glutamate signaling can reverse depressive symptoms, especially in depressed patients with treatment resistance.

Inflammatory cytokines are known to inhibit glutamate reuptake and increase glutamate release from astrocytes, and glutamate antagonists have been shown to block inflammation-induced depressive-like behavior in mice. Moreover, using MRS, data has shown that administration of the inflammatory cytokine interferon (IFN)-alpha significantly increases glutamate in the basal ganglia in association with IFN-alpha-induced anhedonia and psychomotor slowing. In addition, increased inflammation as reflected by peripheral blood C-reactive protein (CRP) is correlated with increased basal ganglia glutamate in association with decreased motivation and psychomotor speed in patients with MDD. Nevertheless, the data to date has been correlational, and whether increased inflammation causes increased glutamate in the basal ganglia, which in turn contributes to behavioral changes in patients with depression has not been established.

To test this hypothesis, investigators plan to determine the cause and effect relationship between increased inflammation and increased CNS glutamate by blocking inflammation in depressed patients with high inflammation (CRP>3mg/L) using the highly specific tumor necrosis factor (TNF) antagonist infliximab (n=30) versus placebo (n=30). In addition, the study team will examine whether changes in basal ganglia glutamate are linked to changes in behaviors related to the basal ganglia including anhedonia and psychomotor retardation.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent
* Primary diagnosis of the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) MDD, current, or Bipolar, depressed type as diagnosed by the SCID-V
* Score of ≥14 on the Quick Inventory of Depressive Symptomatology (QIDS-SR-16) or score ≥ 15 on the Patient Health Questionnaire 9 item (PHQ-9)
* Absence of significant suicidal ideation defined using the Columbia Suicide Severity Rating Scale - Screen Version (CSSRS)
* Off all antidepressant or other psychotropic therapy (e.g. mood stabilizers, antipsychotics, anxiolytics, and sedative hypnotics) for at least 4 weeks prior to the baseline visit (8 weeks for fluoxetine). No patients will be removed from their psychotropic medications for the sole purpose of participating in the study.

Exclusion Criteria:

* Autoimmune disorder (as confirmed by laboratory testing)
* History of tuberculosis (by history or as discovered by chest X-ray, skin testing or blood testing) or high risk of tuberculosis exposure
* Hepatitis B or C infection or human immunodeficiency virus infection (as established by laboratory testing)
* History of fungal infection
* History of recurrent viral or bacterial infections
* History of any type of cancer
* Unstable cardiovascular, endocrinologic, hematologic, hepatic, renal, or neurologic disease (as determined by physical examination and laboratory testing)
* History of any (non-mood-related) psychotic disorder; active psychotic symptoms of any type; antisocial personality disorder as determined by a clinician; substance abuse/dependence within 6 months of study entry (as determined by SCID)
* Active suicidal plan as determined by a score >3 on item #3 on the Hamilton Depression Rating Scale (HAM-D)
* Active eating disorder
* History of a cognitive disorder or ≤28 on the Mini-Mental State Exam
* Pregnancy or lactation
* Women of child bearing potential who are not using a medically accepted means of contraception
* Heterosexual males and their partners who do not agree to practice appropriate birth control
* Known allergy to murine products or other biologic therapies
* Chronic use of non-steroidal anti-inflammatory agents (NSAIDS), glucocorticoid containing medications or statins
* Use of NSAIDS, glucocorticoids, or statins at any time during the study
* Contraindication to MRI
* Previous organ transplant
* History of CNS trauma or active seizure disorder
* Highly treatment resistant depressed patients who score >5 on the Massachusetts General Hospital (MGH) Antidepressant Treatment Response Questionnaire (ATRQ) for current episode

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2019-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew H Miller, MD, Principal Investigator — Emory University; Ebrahim Haroon, MD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Lee Y, Subramaniapillai M, Brietzke E, Mansur RB, Ho RC, Yim SJ, McIntyre RS. Anti-cytokine agents for anhedonia: targeting inflammation and the immune system to treat dimensional disturbances in depression. Ther Adv Psychopharmacol. 2018 Nov 19;8(12):337-348. doi: 10.1177/2045125318791944. eCollection 2018 Dec. PMID 30524702

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Emory University Hospitals and Clinics in Atlanta, Georgia, USA. Participant enrollment began May 15, 2017 and the final follow-up assessment occurred November 27, 2019. The study was suspended in March 2020 during the coronavirus disease 2019 (COVID-19) pandemic. Due to the intervention being an immune suppressant it was not safe to reopen the study to enrollment and the decision was made to terminate the study in March 2023.
Groups:
- Infliximab: Participants randomized to receive one intravenous (IV) infusion of infliximab.
Period: Overall Study
Arm/Group | Infliximab | Placebo
Started | 11 | 11
Completed | 11 | 10
Not Completed | 0 | 1
Not completed — Pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infliximab | Placebo | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (12.8) | 33.3 (9.9) | 38.6 (12.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 6 | 10
  White | 6 | 5 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Central Nervous System (CNS) Glutamate
Description: Left basal ganglia glutamate was measured by magnetic resonance spectroscopy (MRS). Left basal ganglia glutamate tends to be increased during inflammation and is also associated with an increase in depressive symptoms.
Time Frame: Baseline, Day 3, Week 2
Population: Eleven distinct participants in the placebo study arm were examined at least one time point but some had a poor signal scan resulting in non-usable data. One participant in the placebo study arm was removed from the study following the baseline assessment.
Measure: Mean (Standard Deviation); unit: mmol/kg
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 11 | 11
mmol/kg
  Baseline: number analyzed (Participants) | 11 | 10
  Baseline | 7.71 (0.69) | 6.73 (0.64)
  Day 3: number analyzed (Participants) | 11 | 9
  Day 3 | 7.19 (0.93) | 7.81 (0.56)
  Week 2: number analyzed (Participants) | 11 | 9
  Week 2 | 7.41 (0.74) | 7.17 (0.59)

2. Secondary Outcome: Snaith-Hamilton Pleasure Scale - Clinician Administered (SHAPS-C) Score
Description: The SHAPS-C is a 14-item, clinician-administered instrument assessing pleasure response/hedonic experience. Responses are scored as 1 = lots of pleasure, 2 = average/usual pleasure, 3 = some pleasure, and 4 = no pleasure. Total scores range from 14 to 56 where higher scores indicate increasing severity of anhedonia.
Time Frame: Baseline, Day 3, Week 2
Population: One participant in the placebo study arm was removed from the study following the baseline assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 11 | 11
score on a scale
  Baseline | 37.9 (8.2) | 41.7 (6.8)
  Day 3: number analyzed (Participants) | 11 | 10
  Day 3 | 37.2 (9.4) | 39.1 (7.8)
  Week 2: number analyzed (Participants) | 11 | 10
  Week 2 | 32.9 (10.9) | 41.0 (6.9)

3. Secondary Outcome: Mood and Pleasure Scale - Self Report (MAP-SR) Score
Description: The Mood and Pleasure Scale is an 18-item self-report inventory that was created to disentangle state-wise motivational and consummatory components of everyday activities over a 24-hour period. Responses are given on a 5-point Likert scale where 0 = no pleasure/not at all and 4 = extreme pleasure/very often. Total scores range from 0 to 72 and higher scores indicate greater motivation and pleasure during everyday activities.
Time Frame: Baseline, Day 3, Week 2
Population: One participant in the infliximab study arm did not complete this assessment at the Day 3 time point. One participant in the placebo study arm was removed from the study following the baseline assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 11 | 11
score on a scale
  Baseline | 29.3 (3.9) | 23.4 (11.1)
  Day 3: number analyzed (Participants) | 10 | 10
  Day 3 | 29.4 (8.5) | 23.6 (9.5)
  Week 2: number analyzed (Participants) | 11 | 10
  Week 2 | 30.8 (9.6) | 22.6 (10.3)

4. Secondary Outcome: Finger Tapping Task (FTT) Score
Description: The FTT uses a specially adapted tapper that the participant taps as fast as possible using the index finger. The participant is given 5 consecutive 10-second trials for the dominant hands. The finger tapping score is the mean of 5 trials. The FTT is designed to assess subtle motor impairment and is altered in subjects with basal ganglia disorders and lesions. A lower score indicates motor impairment.
Time Frame: Baseline, Day 3, Week 2
Population: One participant in the placebo study arm was removed from the study following the baseline assessment. Some participants did not complete this assessment at the indicated study visits.
Measure: Mean (Standard Deviation); unit: number of taps
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 10 | 10
number of taps
  Baseline | 47.0 (7.8) | 42.4 (8.7)
  Day 3 | 48.4 (7.2) | 46.0 (9.0)
  Week 2: number analyzed (Participants) | 10 | 9
  Week 2 | 46.1 (5.7) | 46.7 (8.0)

5. Secondary Outcome: Digit Symbol Substitution Task (DSST) Score
Description: The DSST is a subtest of the Wechsler Adult Intelligence Scale (WAIS) and consists of rows of blank squares, each printed with a randomly assigned number. The test involves graphomotor speed, visual scanning and memory, with about half of the variance being accounted for by graphomotor speed, a third by visual scanning and 4-5% by memory. Performance on the DSST has been found to correlate with subcortical atrophy in disorders involving basal ganglia.The DSST is scored as the number of correct responses in 120 seconds, with higher scores indicating better performance.
Time Frame: Baseline, Day 3, Week 2
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: correct responses
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 10 | 10
correct responses
  Baseline | 55.5 (15.0) | 60.0 (16.6)
  Day 3 | 63.8 (16.4) | 67.9 (21.1)
  Week 2: number analyzed (Participants) | 10 | 9
  Week 2 | 64.2 (17.4) | 62.9 (15.2)

6. Secondary Outcome: Trails Making Test A (TMT-A) Score
Description: The scale measures cognitive processing speed using a series of non-sequentially arranged numbers where the participant is asked to sequentially track the numbers occurring to numerical order as quickly as possible. The score is the time time it takes to complete the task, measured in seconds. A longer time to finish may indicate cognitive impairment.
Time Frame: Baseline, Day 3, Week 2
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 10 | 11
seconds
  Baseline | 28.4 (7.6) | 24.9 (7.9)
  Day 3: number analyzed (Participants) | 10 | 10
  Day 3 | 23.5 (8.0) | 22.4 (8.2)
  Week 2: number analyzed (Participants) | 10 | 10
  Week 2 | 19.4 (3.6) | 20.9 (7.6)

7. Secondary Outcome: Multidimensional Fatigue Inventory (MFI) Score
Description: The Multidimensional Fatigue Inventory (MFI) is a 20-item self-report instrument designed to measure motivation and fatigue, covering the dimensions of General Fatigue, Physical Fatigue, Mental Fatigue, Reduced Motivation and Reduced Activity. Participants respond to fatigue related statements using a 5-point scale where 1 = "yes, that is true" and 5 = "no, that is not true". Total scores range from 20 to 100 and higher scores indicate greater fatigue.
Time Frame: Baseline, Day 3, Week 2
Population: One participant in the placebo study arm was removed from the study following the baseline assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 11 | 11
score on a scale
  Baseline | 77.3 (11.8) | 75.8 (11.9)
  Day 3: number analyzed (Participants) | 11 | 10
  Day 3 | 71.4 (14.4) | 72.8 (16.1)
  Week 2: number analyzed (Participants) | 11 | 10
  Week 2 | 72.3 (15.1) | 71.6 (16.4)

8. Secondary Outcome: Inventory of Depressive Symptoms-Clinician Rating (IDS-SR) Score
Description: The Inventory of Depressive Symptomatology-Self-Report (IDS-SR) is a 30-item self-report instrument designed to measure symptom constructs consistent with current Diagnostic and Statistical Manual of Mental Disorders (DSM) nosology and that has been widely used as a self-report outcome measure of depression. Participants complete 28 of the 30 items, depending on if they experienced an increase or decrease in appetite and weight. Each item is scored on a 4-point scale where 0 means that the symptom is absent and 3 means that the symptom is very strongly felt. Total scores can range between 0 and 84 and higher scores indicate more severe symptoms of depression.
Time Frame: Baseline, Day 3, Week 2
Population: One participant in the placebo study arm was removed from the study following the baseline assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 11 | 11
score on a scale
  Baseline | 30.7 (8.2) | 39.7 (14.6)
  Day 3: number analyzed (Participants) | 11 | 10
  Day 3 | 26.4 (12.6) | 32.6 (14.6)
  Week 2: number analyzed (Participants) | 11 | 10
  Week 2 | 23.5 (10.9) | 32.7 (12.3)

9. Secondary Outcome: Plasma Concentrations of High-sensitivity C-reactive Protein (Hs-CRP)
Description: This study collected blood samples to assess inflammatory markers. Increases in hsCRP are seen when inflammation is present.
Time Frame: Baseline, Day 3, Week 2
Population: One participant in the placebo study arm was removed from the study following the baseline assessment. Samples were not obtained for one participant in the Infliximab group at Baseline and for one participant in the Placebo group at Week 2.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 11 | 11
mg/L
  Baseline: number analyzed (Participants) | 10 | 11
  Baseline | 5.70 (5.74) | 5.85 (7.54)
  Day 3: number analyzed (Participants) | 11 | 10
  Day 3 | 4.74 (5.58) | 6.32 (5.71)
  Week 2: number analyzed (Participants) | 11 | 9
  Week 2 | 9.02 (14.60) | 4.97 (4.99)

10. Secondary Outcome: Plasma Concentrations of Tumor Necrosis Factor Alpha (TNF-α)
Description: This study collected blood samples to assess inflammatory markers. TNF-α is elevated in patients experiencing inflammation and a decrease in serum TNF-α is an indication of effective treatment.
Time Frame: Baseline, Day 3, Week 2
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 11 | 11
pg/mL
  Baseline: number analyzed (Participants) | 10 | 11
  Baseline | 3.78 (1.45) | 4.50 (1.75)
  Day 3: number analyzed (Participants) | 11 | 10
  Day 3 | 1.69 (1.13) | 4.12 (1.99)
  Week 2: number analyzed (Participants) | 11 | 9
  Week 2 | 2.69 (1.21) | 4.65 (2.20)

11. Secondary Outcome: Plasma Concentrations of Tumor Necrosis Factor (TNF) Receptor 2 (TNFR2)
Description: This study collected blood samples to assess inflammatory markers. TNFR2 has proinflammatory effects and has strong anti-inflammatory activities.
Time Frame: Baseline, Day 3, Week 2
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 11 | 11
pg/mL
  Baseline: number analyzed (Participants) | 10 | 11
  Baseline | 1610.66 (647.10) | 1956.91 (698.70)
  Day 3: number analyzed (Participants) | 11 | 10
  Day 3 | 1451.14 (589.90) | 2028.00 (774.03)
  Week 2: number analyzed (Participants) | 11 | 9
  Week 2 | 1774.36 (1042.49) | 2049.67 (814.24)

12. Secondary Outcome: Plasma Concentrations of Interleukin-1 Receptor Antagonist (IL-1Ra)
Description: This study collected blood samples to assess inflammatory markers. IL-1Ra is an anti-inflammatory protein secreted by immune cells, epithelial cells, and adipocytes.
Time Frame: Baseline, Day 3, Week 2
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 11 | 11
pg/mL
  Baseline: number analyzed (Participants) | 10 | 11
  Baseline | 463.53 (171.46) | 394.40 (174.07)
  Day 3: number analyzed (Participants) | 11 | 10
  Day 3 | 482.49 (279.85) | 404.43 (169.55)
  Week 2: number analyzed (Participants) | 11 | 9
  Week 2 | 519.32 (296.09) | 440.34 (226.75)

13. Secondary Outcome: Plasma Concentrations of IL-6
Description: This study collected blood samples to assess inflammatory markers. IL-6 is a proinflammatory cytokine that is elevated during times of inflammation, infection, illness, and in patients with mood disorders. IL-6 is not present or is low in healthy individuals and exact reference ranges vary by lab, with an example normal reference range of 0.31 to 5.00 picograms per milliliter (pg/mL).
Time Frame: Baseline, Day 3, Week 2
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 11 | 11
pg/mL
  Baseline: number analyzed (Participants) | 10 | 11
  Baseline | 0.75 (0.48) | 0.91 (0.33)
  Day 3: number analyzed (Participants) | 11 | 10
  Day 3 | 0.62 (0.36) | 0.98 (0.63)
  Week 2: number analyzed (Participants) | 11 | 9
  Week 2 | 0.58 (0.22) | 1.00 (0.59)

14. Secondary Outcome: Plasma Concentrations of Soluble IL-6 Receptor (sIL-6R)
Description: This study collected blood samples to assess inflammatory markers. Working with the pro-inflammatory cytokine IL-6, sIL-6R regulates pro-inflammatory reactions.
Time Frame: Baseline, Day 3, Week 2
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 11 | 11
pg/mL
  Baseline: number analyzed (Participants) | 10 | 11
  Baseline | 30539.70 (5791.88) | 31108.64 (8243.70)
  Day 3: number analyzed (Participants) | 11 | 10
  Day 3 | 32963.18 (6499.08) | 30732.30 (7834.47)
  Week 2: number analyzed (Participants) | 11 | 9
  Week 2 | 31062.73 (7594.65) | 32156.56 (7290.96)

15. Post Hoc Outcome: Plasma Concentrations of IL-1 Beta
Description: This study collected blood samples to assess inflammatory markers. IL-1 Beta is a mediator of the inflammatory response and increased levels are present with a stronger inflammatory stimulus.
Time Frame: Baseline, Day 3, Week 2
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 11 | 11
pg/mL
  Baseline: number analyzed (Participants) | 10 | 11
  Baseline | 0.24 (0.0) | 0.25 (0.06)
  Day 3: number analyzed (Participants) | 11 | 10
  Day 3 | 0.24 (0.04) | 0.24 (0.11)
  Week 2: number analyzed (Participants) | 11 | 9
  Week 2 | 0.25 (0.06) | 0.48 (0.68)

16. Post Hoc Outcome: Plasma Concentrations of Monocyte Chemoattractant Protein-1 (MCP-1)
Description: This study collected blood samples to assess inflammatory markers. Elevated levels of MCP-1 are present with several disease conditions including neuroinflammatory diseases.
Time Frame: Baseline, Day 3, Week 2
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 11 | 11
pg/mL
  Baseline: number analyzed (Participants) | 10 | 11
  Baseline | 122.59 (18.72) | 121.70 (31.92)
  Day 3: number analyzed (Participants) | 11 | 10
  Day 3 | 123.51 (28.42) | 124.32 (25.55)
  Week 2: number analyzed (Participants) | 11 | 9
  Week 2 | 117.96 (15.81) | 128.50 (24.41)

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the baseline assessment and continued through the final assessment at Week 2.
Arm/Group | Infliximab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/11 | 0/11
Other Adverse Events (participants affected / at risk) | 6/11 | 8/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infliximab (N=11) | Placebo (N=11)
Serotonin syndrome after study completion and after receiving escitalopram (Product Issues) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infliximab (N=11) | Placebo (N=11)
Venipuncture site bruise (Surgical and medical procedures) | 1 | 4
Venipuncture stie pain (Surgical and medical procedures) | 1 | 2
Infusion site pain (Surgical and medical procedures) | 1 | 0
Vascular access failure (Surgical and medical procedures) | 1 | 0
Adhesive reaction (Surgical and medical procedures) | 1 | 0
Fatigue (General disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Shoulder tightness (Musculoskeletal and connective tissue disorders) | 1 | 0
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (General disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 1 | 0
Lightheadedness (General disorders) | 1 | 1
Dizziness (General disorders) | 0 | 2
Puncture site pain (Surgical and medical procedures) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
External ear pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Parethesia (Nervous system disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Upper respiratory infection (Infections and infestations) | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Increased appetite (General disorders) | 0 | 1
Infusion site irritation (Surgical and medical procedures) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-14): https://cdn.clinicaltrials.gov/large-docs/43/NCT03004443/Prot_SAP_001.pdf
  • Informed Consent Form (2019-10-23): https://cdn.clinicaltrials.gov/large-docs/43/NCT03004443/ICF_000.pdf